CLINICAL TRIAL: NCT05603117
Title: A Single Case Experimental Design Investigating CISBAR Intervention for Improving Social Communication After ABI
Brief Title: CISBAR Intervention for Social Communication After ABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Principal Investigator, Heidi Iwashita, Doctoral candidate, University of Oregon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12292020.033
Record Dates: First submitted 2022-08-29; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants received a behavioral intervention, CISBAR, via zoom sessions.
  Interventions: Behavioral: Collaborative Interpersonal Strategy Building with Audio Reflection (CISBAR)

INTERVENTIONS:
Behavioral: Collaborative Interpersonal Strategy Building with Audio Reflection (CISBAR) — CISBAR incorporates collaborative, individualized goal-setting, metacognitive strategy training, audio feedback, reflection, and practice, integrated with the Conversational Rating System for ABI (CoRS-ABI) and adding a new method for selecting individualized and equivalently challenging conversation practice topics.

SUMMARY:
This was the first trial of a new intervention, Collaborative Interpersonal Strategy Building with Audio Reflection (CISBAR), for improving social communication in adults following brain injury. When developing CISBAR, I aimed to provide speech-language pathologists (SLPs) with an integrated package for goal-setting and treatment of social communication after ABI by combining motivational interviewing and goal attainment scaling with evidence-based treatment elements drawn from social cognitive and conversational coaching approaches. To elicit the targeted communication behaviors, CISBAR adds a new system of selecting equivalent conversation topics. To foster self-awareness and reflection, CISBAR incorporates the Conversational Rating System for ABI (CoRS-ABI). I used a single-case experimental, multiple-probe design across participants to evaluate CISBAR.

DETAILED DESCRIPTION:
This was the first trial of a new intervention, Collaborative Interpersonal Strategy Building with Audio Reflection (CISBAR). CISBAR aims to provide speech-language pathologists (SLPs) with an integrated package for goal-setting and treatment of social communication after ABI by combining motivational interviewing and goal attainment scaling with evidence-based treatment elements drawn from social cognitive and conversational coaching approaches. To elicit the targeted communication behaviors, CISBAR adds a new system of selecting equivalent conversation topics. To foster self-awareness and reflection, CISBAR incorporates the Conversational Rating System for ABI (CoRS-ABI).

ELIGIBILITY:
Inclusion Criteria Separate sets of inclusion criteria were used for the primary participants and the ECPs.

Primary Participant Inclusion Criteria:

1. Adults aged 18-80 with reported ABI after age 16.
2. Access to a computer, mobile phone, or tablet with Internet connectivity and a camera in order to allow participation in Zoom sessions; participation may require assistance of everyday communication partner (ECP)
3. Memory ability sufficient to allow meaningful participation in therapy and retention of skills with practice, as determined by the clinician in the initial screening interview with participant and everyday communication partner.
4. Reported ABI greater than eight months prior with hospitalization of at least one day resulting in changes in cognitive communication
5. Able to identify an ECP (i.e., a close friend or family member with whom the participant talks at least once per week), who is willing to participate in each session and whom the primary participant endorses as supportive.
6. Participant and ECP report current challenges in social communication characterized by verbosity (or limited speech), tangentiality and/or difficulty taking the perspective of others which were not apparent before the ABI
7. Participant and the ECP both indicate willingness to work on measurable social communication behaviors (specifically interruption, wordiness, limited speech, or perspective taking) using the present intervention. Specifically, both the participant and ECP must score midway or above on the Motivational Interviewing (MI) rulers of confidence in change and importance of change (Miller & Rollnick, 2013; described below in the Initial Intake section).
8. Participants must be able to participate in therapy without significant barriers to treatment posed by severe depression or other mental health issues, as determined by the screening interview with the ECP and primary participant, and results of The Depression Anxiety Stress Scales-21 (DASS-21; Lovibond & Lovibond, 1995).

ECP Inclusion Criteria:

1. Nominated by the primary participant as a person who talks with the primary participant regularly (at least once per week).
2. Endorsed by the primary participant as being supportive.
3. Willing to participate in each session with the primary participant.
4. Indicates readiness to support the participant in working on a communication goal by scoring at least midway on the Motivational Interviewing (MI) rulers of confidence in change and importance of change (Miller & Rollnick, 2013; described below in the Initial Intake section).
5. Demonstrated satisfactory supportiveness in communication as indicated by scores of at least 2 out of 4 on the Measure of Skill in Supported Conversation (MSC) scales of the adapted Kagan Scales (Togher et al., 2010), indicating a basic level of skill in acknowledging competence and revealing competence in the person with ABI, after a short training in supportive communication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Number of interruptions | 6-7 minutes
  number of times the participant interrupted their partner
Average duration of speaking turn | 6-7 minutes
  average number of seconds of speaking turn in conversation with partner

CONTACTS AND LOCATIONS:
Overall Officials: McKay M Sohlberg, PhD, Study Chair — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
with additional consent given by participants under the oversight of the IRB at Eastern Washington University (EWU), videorecorded intervention sessions may be made available to student researchers for further research.
Supporting Information: Study Protocol, ICF
Time Frame: Two participants have given additional consent for their data to be used by a research student for further analysis. The time frame of access is under the oversight of the EWU IRB according to the protocol of a separate IRB-approved study.

DOCUMENTS (2):
  • Informed Consent Form: version for participants with history of brain injury (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT05603117/ICF_000.pdf
  • Informed Consent Form: version for everyday communication partner (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT05603117/ICF_001.pdf